CLINICAL TRIAL: NCT06204523
Title: Prospective Validation of a DNA Damage Repair-Hippo Pathway Signature in Patients With Advanced Gastric Cancer
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Regina Elena Cancer Institute (Other)
Collaborators: Azienda Sanitaria Locale n. 2 - Lanciano Vasto Chieti (Other); Campus Bio-Medico University (Other); Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other); Azienda Ospedaliera "Sant'Andrea" (Other); University of Roma La Sapienza (Other); Azienda Ospedaliero Universitaria Policlinico Modena (Other)
Responsible Party: Sponsor
Other Study IDs: RS1043/18
Record Dates: First submitted 2023-03-28; First posted 2024-01-12 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: DNA Damage; Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Popolation
  Interventions: Diagnostic Test: investigated biomarkers regarding the efficacy of first-line chemotherapy

INTERVENTIONS:
Diagnostic Test: investigated biomarkers regarding the efficacy of first-line chemotherapy — The present study was designed to generate solid evidence on the predictivity of the investigated biomarkers regarding the efficacy of first-line chemotherapy in patients with GC

SUMMARY:
We envisioned a scenario where the interaction between the ATM-Chk2/ATR-Chk1 pathways and Hippo enables GC cells to overcome chemotherapy-induced death stimuli. First, ATM-Chk2 and ATR-Chk1 were found to be activated across all the GC molecular subtypes. Moreover, a number of genes associated with their basal activation are recurrently mutated or amplified.

Thus, we retrospectively characterized a cohort of GC patients treated with first-line therapy for DDR- and Hippo-related markers, identifying a signature predicting inferior PFS and OS. This exploratory analysis provided the necessary information (frequency of candidate biomarkers and effect difference between groups) for a prospective study with validation purposes, which is the main goal of this trial.

DETAILED DESCRIPTION:
This prospective, multicenter, non-interventional trial is designed for prospectively validating the DDR-Hippo signature as a predictor of inferior PFS in patients with inoperable locally advanced or metastatic GC receiving first-line therapy. Patients will be evaluated for response to chemotherapy every two cycles by current RECIST criteria. PFS will be defined as the time elapsing between the initiation of chemotherapy until objective tumor progression or death, and OS as the time elapsing between the initiation of chemotherapy until death from any cause. All molecular analyses will be centralized at the coordinating center. Investigators performing molecular analyses will be masked to clinical outcomes. Centralized radiological review is planned. The study will be conducted in accordance with the Declaration of Helsinki and adheres to the REMARK criteria.

The second task is designed for exploring genetic events functionally related to the DDR and Hippo pathways that may modify the predictive significance of the signature. These genes are schematically clustered on the basis of the expected alteration in: i) Mutated genes (cluster 1) to be evaluated by targeted DNA-Seq and amplified genes (cluster 2) to be evaluated by FISH/CISH. Cluster 1 includes TP53 (defective cell cycle progression and apoptotic response, aberrant TAZ/YAP-mediated transcription), KRAS (oncogene-induced replication stress and activation of cell cycle checkpoints to avoid apoptosis and senescence), BRCA1 and BRCA2 (defective homologous recombination repair), ARID1A, ATR and ATM (altered ATM/ATR-initiated DNA repair), RHOA (G-protein coupled receptor-mediated activation of TAZ/YAP), CTNNB1, APC and FBXW7 (Wnt-mediated control of TAZ/YAP). Cluster 2 encompasses MYC and KRAS (oncogene-induced replication stress), CCNE1, CCND1 and CDK6 (dysfunctional G1-S transition requiring compensatory activation of intra-S and G2/M checkpoints).

The present study is designed to generate prospective evidence on the ability of the investigated biomarkers to predict the efficacy of first-line chemotherapy in GC patients. The identification of patients who derive marginal benefit from chemotherapy holds the potential to expedite a wave of interventional trials with agents targeting the DDR-Hippo network (e.g. PARP inhibitors and ATR-Chk1 and ATM-Chk2 inhibitors), as well as to delineate the target population for studies with other compounds, such as immune checkpoint inhibitors. Overall, the experimental approach we propose is expected to culminate in the generation of a new tool to be used on a routine basis.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years;
* Histologic diagnosis of locally advanced or metastatic gastric carcinoma (GC) or gastroesophageal junction carcinoma (EJC);
* Biological material adequate for molecular analysis to be performed, taken (at surgery or by biopsy) prior to the administration of any anti-tumor treatment (chemotherapy and/or radiotherapy);
* ECOG PS 0-2;
* Adequate hematologic, hepatic, and renal function;
* Measurable disease according to RECIST criteria;
* Written informed consent.

Exclusion Criteria:

* Previous chemotherapy for metastatic disease;
* Comorbidities not controlled with appropriate medical therapy;
* Brain metastasis;
* Patient unable to give adequate consent for the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with inoperable locally advanced or metastatic GC who are candidates for first-line chemotherapy treatment and meet the following criteria will be included in the study
Sampling Method: Non-Probability Sample
Enrollment: 167 (Estimated)
Dates: Start 2018-10-26 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2024-08-30 (Estimated)

PRIMARY OUTCOMES:
Identify new biomarkers that predict the activity of first-line chemotherapy, in order to achieve better patient selection. | Three years
  Computational enrichment analysis will be carried out to test whether tumors of patients with shorter PFS contain a higher-than-randomly-expected representation of a specific pathway/function. Special emphasis will be placed on, but not limited to, the DDR-Hippo-Wnt pathways. For multiple hypothesis testing a Benjamini-Hochberg False Discovery Rate correction will be applied (<5%). For clinical data analysis, the Pearson's Chi-squared test of independence (2-tailed) and the Pearson's correlation coefficient will be used to assess the relationships between categorical and continuous variables, respectively.
Identify additional genetic events molecularly linked to the DDR-Hippo signature and potentially improve its predictive ability. | Three years
  RNA and DNA will be extracted from 5µm FFPE tissue sections using the AllPrep DNA/RNA FFPE kit (Qiagen). Libraries for RNA-Seq will be prepared using the TruSeq Stranded Total RNA kit with an initial ribosomal depletion step (Illumina). Targeted DNA-Sequencing will be conducted by designing a custom amplicon panel with DesignStudio and employing the TruSeq Custom Amplicon Low Input Kit (Illumina). RNA will be analyzed with our cloud pipeline (RAP, available at https://bioinformatics.cineca.it/rap/) that employs the Tuxedo Suite (Tophat, Cufflinks, Cuffdiff).
  For DNA analysis, applications available on Basespace (Illumina) will be used. Sequencing will be performed on our NextSeq500
Investigate pathways of interest at a deeper level, as well as identify other potential pathways/functions impacting clinical outcomes. | Three years
  Clinical, pathological and molecular variables will be tested in univariate Cox analysis. A multivariate Cox proportional hazard model for PFS will be build with variables testing significant at the univariate assessment, and the related estimates reported as HR and 95%CI.

CONTACTS AND LOCATIONS:
Locations (1):
- "Regina Elena" National Cancer Institute, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided